CLINICAL TRIAL: NCT05642247
Title: Quantify the Value of Transmural Inflammation in the Treatment of Crohn's Disease With Ustekinumab:an Analysis Based on Imaging Science
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022ZSLYEC-317
Record Dates: First submitted 2022-08-30; First posted 2022-12-08 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Biologics
Keywords: Crohn Disease; Biologics
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CD patients who received Ustekinumab treatment: 1. Inpatients with Crohn's disease diagnosed in the Sixth Affiliated Hospital of Sun Yat-Sen University from January 2020 to June 2022. 2.The patients were treated with Ustekinumab and followed up regularly for 20 weeks. 3. Complete pre-treatment cross-sectional imaging data (CTE/MRE and US)

SUMMARY:
Crohn's disease(CD),a type of inflammatory bowel disease(IBD), is a chronic intestinal recurrent inflammatory disease involving the entire digestive tract. And Ustekinumab, a monoclonal antibody against the p40 subunit of interleukin-12 and interleukin-23, is a newly targeted drug approved for the treatment of Crohn's disease in recent years.Based on the high-throughput imaging characteristic analysis technique, this study quantitatively analyzed the transmural inflammation of Crohn's disease, and discussed its prognostic value in the treatment of Ustekinumab, and further analyzed the increment of its relative clinical index.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with Crohn's disease diagnosed in the IBD center of Sixth Affiliated Hospital of Sun Yat-Sen University from January 2020 to June 2022
* Treated with Ustekinumab and followed up regularly for 20 weeks
* Complete pre-treatment cross-sectional imaging data (CTE/MRE and US)

Exclusion Criteria:

* The diagnosis is not clear
* Under the age of 18
* Lack of endoscopic and pathological data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: January 2020 to June 2022 CD patients in the IBD center of Sixth Affiliated Hospital of Sun Yat-Sen University, who were treated with Ustekinumab.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
endoscopic remission rate at 12 months | 12 months after first intervention administration
  endoscopic remission rate at 12 months
normalization rate of serum biomarker at 12 months | 12 months after first intervention administration
  normalization rate of serum biomarker at 12 months
clinical remission rate at 12 months | 12 months after first intervention administration
  clinical remission rate at 12 months
clinical response rate at 12 months | 12 months after first intervention administration
  clinical response rate at 12 months
endoscopic response rate at 12 months | 12 months after first intervention administration
  endoscopic response rate at 12 months
life quality changes at 12 months | 12 months after first intervention administration
  life quality evaluated by CDAI (Crohn's Disease Activity Index) at 12 months
endoscopic remission rate after induction therapy | 16 or 20 weeks after first intervention administration
  endoscopic remission rate after induction therapy
normalization rate of serum biomarker after induction therapy | 16 or 20 weeks after first intervention administration
  normalization rate of serum biomarker after induction therapy
clinical remission rate after induction therapy | 16 or 20 weeks after first intervention administration
  clinical remission rate after induction therapy
clinical response rate after induction therapy | 16 or 20 weeks after first intervention administration
  clinical response rate after induction therapy
endoscopic response rate after induction therapy | 16 or 20 weeks after first intervention administration
  endoscopic response rate after induction therapy
life quality changes after induction therapy | 16 or 20 weeks after first intervention administration
  life quality evaluated by CDAI (Crohn's Disease Activity Index) after induction therapy

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China